CLINICAL TRIAL: NCT03122873
Title: Quantitation of McArdle's Sign and Evaluation of Specificity for Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian G. Weinshenker, M.D., PI, Mayo Clinic
Other Study IDs: 15-009122
Record Dates: First submitted 2017-04-06; First posted 2017-04-21 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Myelopathy of any cause: Male or female 18 years or older with myelopathy and detectable finger extension weakness due to 1) prototypic multiple sclerosis (N=50) 2) other etiologies of myelopathy (N=50), including other inflammatory conditions (e.g. idiopathic transverse myelitis, neuromyelitis optica, acute disseminated encephalomyelitis, sarcoidosis) or other etiologies (compression, vascular disorders, degenerative disorders, neoplasms).
- Peripheral neuropathy: Male or female 18 years or older with C7 radiculopathy, radial neuropathy, plexopathy, peripheral neuropathy, who have detectable finger extension weakness.
- Healthy Controls: Male and female 18 year or older with no finger extension weakness and no known neurological conditions.

SUMMARY:
The study is designed to quantitate McArdle's sign, an increase in measurable weakness with neck flexion described in patients with multiple sclerosis, and to determine whether it is or is not specific for multiple sclerosis.

DETAILED DESCRIPTION:
Finger strength will be measure using a torque-measuring device designed to quantitate finger extension strength. The device was designed for point of treatment use, patient safety and portability. Strength will be measured in 5 paired trials, first with neck extended and then with neck flexed. Two protocols will be evaluated, one testing isometric strength against a fixed resistance and the second testing strength against dynamic resistance. McArdle's sign is the difference between strength with neck extension and strength with neck flexion.

The data will be digitally registered and dynamic neck position will be recorded electronically in real time. Graphs of dynamic changes in torque versus neck position will be generated and superimposed. Strength will be quantitated using Matlab software.

Consecutive patients with myelopathy of any cause with detectable finger extensor weakness will be studied, either due to MS or due to other cause of myelopathy (other inflammatory, vascular, compressive, neoplastic and other). Additionally, normal controls will be studied as will patients with finger extension weakness due to peripheral nerve lesions.

ELIGIBILITY:
Inclusion Criteria:

* Myelopathy of any cause with finger extension weakness
* Patients with peripheral neuropathy with finger extension weakness
* Healthy controls

Exclusion Criteria:

* Pregnant subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with myelopathy of any cause and peripheral neuropathy who have detectable finger extension weakness.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in quantitative measure of strength between extended positions of the neck and fully flexed position of the neck (McArdle's sign) | through study completion, an average of 1 year
  Comparison of means and medians of the difference in strength in the fully extended and fully flexed positions ("McArdle's sign") measured using a torque measurement device between multiple sclerosis versus other myelopathy and between multiple sclerosis and normal controls; measurements are done in 5 successive trials of extension and flexion and the mean percentage difference between extension and flexion of the last 4 trials is averaged to calculated the McArdle's sign; the goal is to determine whether there is a specific level of McArdle sign that is diagnostic for MS using receiver operator curve method.

SECONDARY OUTCOMES:
Relative sensitivity of clinical versus instrument-based detection of McArdle's sign. | through study completion, an average of 1 year
  Compare the clinical detection of the sign by the referring clinician and technician compared to the device-determined McArdle's sign

CONTACTS AND LOCATIONS:
Overall Officials: Brian Weinshenker, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Savoldi F, Nasr Z, Hu W, Schilaty ND, Delgado AM, Mandrekar J, Kaufman KR, Berglund L, Weinshenker BG. McArdle Sign: A Specific Sign of Multiple Sclerosis. Mayo Clin Proc. 2019 Aug;94(8):1427-1435. doi: 10.1016/j.mayocp.2019.01.047. Epub 2019 Jul 11. PMID 31303427